CLINICAL TRIAL: NCT07055516
Title: A Phase 2a Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Efficacy and Safety of NT-0796 as an Adjunct to a Reduced Calorie Diet and Increased Physical Activity in Obese Participants With/Without Type 2 Diabetes
Brief Title: Evaluate the Efficacy and Safety of NT-0796 in Participants With Obesity With or Without Type 2 Diabetes Mellitus
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: NodThera Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NT-0796-P004
Record Dates: First submitted 2025-05-30; First posted 2025-07-09 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: Obesity and Type 2 Diabetes
Keywords: NLRP3; T2DM; NT-0796; Obesity; RESOLVE-1
MeSH Terms: conditions — Obesity; Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Twice daily orally administered NT-0796 capsule (Experimental): Participants will receive study medication twice daily orally for up to 24 weeks, containing NT-0796 twice daily
  Interventions: Drug: NT-0796
- Once daily orally administered NT-0796 capsules and placebo second daily dose (Experimental): Participants will receive study medication twice daily orally for up to 24 weeks, containing NT-0796 once daily, with once daily placebo
  Interventions: Drug: NT-0796; Drug: Placebo
- Placebo orally administered capsule (Placebo Comparator): Participants will receive placebo twice daily orally for up to 24 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: NT-0796 — Orally administered capsules
  Arms: Once daily orally administered NT-0796 capsules and placebo second daily dose; Twice daily orally administered NT-0796 capsule
Drug: Placebo — Orally administered capsules
  Arms: Once daily orally administered NT-0796 capsules and placebo second daily dose; Placebo orally administered capsule

SUMMARY:
A Phase 2a Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Efficacy and Safety of NT-0796 as an Adjunct to a Reduced Calorie Diet and Increased Physical Activity in Obese Participants With/Without Type 2 Diabetes over a 6 months treatment period.

DETAILED DESCRIPTION:
Potential participants will be screened within 28 days prior to baseline (Day 1), and eligible participants will be randomized 1:1:1 within each strata (T2DM or non-T2DM) to either NT-0796 twice daily (BID), NT-0796 once daily (QD) or placebo (BID). Study drug will be administered orally. Following 24 weeks of active treatment, participants will enter a 4-week safety follow-up before being discharged from the study. The primary endpoint of the study will be percentage weight change from baseline, the key-secondary endpoint will be change in HbA1c from baseline in the T2DM stratum, while secondary endpoints include DEXA scans, a variety of other relevant biometric measures as well as biomarkers. Pharmacokinetic, safety and tolerability as well as suicidality will also be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged 18 to 75 years (inclusive) at screening who have signed informed consent and are willing and able to comply with the study protocol.
* Have a BMI of ≥30.0 kilogram/square meter (kg/m2) and <40.0 kg/m2. (BMI values should be calculated to one decimal point precision and then assessed in terms of the required range.)
* History of at least one self-reported unsuccessful dietary effort to lose body weight.
* Group 1: Have a diagnosis of T2DM, with HbA1c ≥6.5% (48 mmol/mol) but < 10% (86 mmol/mol) (measured at central lab during screening) and are on stable treatment for T2DM for at least 90 days prior to screening.
* Group 2: No diagnosis or signs/symptoms of T2DM and HbA1c < 6.5% (48 mmol/mol), measured at the central lab during screening.

Exclusion Criteria:

* T1DM, or a history of ketoacidosis, or hyperosmolar state/coma requiring hospitalization at any time prior to screening.
* Have had 1 or more episode(s) of severe hypoglycemia in the 6 months prior to screening (Level 3 ADA 2025) defined as a severe event characterized by altered mental and/or physical status requiring assistance for treatment of hypoglycemia irrespective of glucose level, or has a history of hypoglycemia unawareness or poor recognition of hypoglycemic symptoms. Any participant that the investigator feels will not be able to communicate an understanding of hypoglycemic symptoms and the appropriate treatment of hypoglycemia should also be excluded.
* History of stroke with residual neurological deficit within 2 years or transient ischemic attack within 6 months prior to Day 1.
* History of acute coronary syndrome (ACS) including unstable angina, acute myocardial infarction (both ST segment elevation and non-ST segment elevation) within 6 months prior to Day 1.
* Diagnosis of congestive heart failure (CHF) or clinical evidence suggesting CHF including history of orthopnea, exertional dyspnea, pedal edema, pulmonary rales, hepatosplenomegaly or cardiomegaly at the discretion of the Principal Investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 162 (Estimated)
Dates: Start 2025-05-08 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Change in body weight in participants with obesity with and without T2DM | Baseline to Week 24

SECONDARY OUTCOMES:
HbA1c in participants with T2DM | Baseline to Week 24
Change in body weight in participants with obesity with and without T2DM | Baseline to week 4, 8, 12, 16 and 20
Change in waist circumference in participants with obesity with and without T2DM | Baseline to week 4, 8, 12, 16, 20 and 24
Change in waist/height ratio in participants with obesity with and without T2DM | Baseline to week 4, 8, 12, 16, 20 and 24
Incidence of body weight loss ≥5% in participants with obesity with and without T2DM | Baseline to Week 24
Incidence of body weight loss ≥10% in participants with obesity with and without T2DM | Baseline to Week 24
Incidence of body weight loss ≥15% in participants with obesity with and without T2DM | Baseline to Week 24
Change in metabolic biomarker in participants with and without T2DM | Baseline to Week 24
Change in lean mass as measured by Dual-energy Xray absorptiometry (DEXA) in participants with obesity with and without T2DM | Baseline to Week 24
Change in bone mineral density as measured by Dual-energy Xray absorptiometry (DEXA) in participants with obesity with and without T2DM | Baseline to Week 24
Incidence of adverse events in participants with obesity with and without T2DM | Baseline to Week 28
Pharmacokinetics (PK); Area Under the Concentration vs. Time curve of NT0796 in participants with obesity with and without T2DM | Baseline to Week 24
PK; Maximum Plasma Concentration (Cmax) of NT0796 in participants with obesity with and without T2DM | Baseline to Week 24

CONTACTS AND LOCATIONS:
Locations (11):
- United States (11):
  - Investigative site, Mesa, Arizona
  - Investigative site, Los Angeles, California
  - Investigative site, Cooper City, Florida
  - Investigative Site, Hialeah, Florida
  - Investigative Site, Jacksonville, Florida
  - Investigative Site, Miami, Florida
  - Investigative Site, Port Orange, Florida
  - Investigative Sites, Marrero, Louisiana
  - Investigative Site, Columbus, Ohio
  - Investigative Site, Dallas, Texas
  - Investigative Site, Manassas, Virginia